CLINICAL TRIAL: NCT02539641
Title: Bariatric Procedures and Changes in Incretins and Gastric Emptying
Acronym: BIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL50111.091.14
Record Dates: First submitted 2015-08-20; First posted 2015-09-03 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Good responder RYGB (Other): Good responders after Roux-en-Y gastric bypass (RYGB). EWL > 50%. Interventions: Gastric emptying scintigraphy and Determination of gut hormones.
  Interventions: Radiation: Gastric emptying scintigraphy; Other: Determination of gut hormones
- Bad responder RYGB (Other): Bad responders after Roux-en-Y gastric bypass (RYGB). EWL < 50% Interventions: Gastric emptying scintigraphy and Determination of gut hormones.
  Interventions: Radiation: Gastric emptying scintigraphy; Other: Determination of gut hormones
- Good responder SG (Other): Good responders after sleeve gastrectomy (SG). EWL > 50% Interventions: Gastric emptying scintigraphy and Determination of gut hormones.
  Interventions: Radiation: Gastric emptying scintigraphy; Other: Determination of gut hormones
- Bad responder SG (Other): Bad responders after sleeve gastrectomy (SG). EWL < 50% Interventions: Gastric emptying scintigraphy and Determination of gut hormones.
  Interventions: Radiation: Gastric emptying scintigraphy; Other: Determination of gut hormones
- Duodenal-jejunal bypass liner (Other): Patients who will have a duodenal-jejunal bypass liner (DJBL) Intervention: Gastric emptying scintigraphy before and after implantation of DJBL
  Interventions: Radiation: Gastric emptying scintigraphy

INTERVENTIONS:
Radiation: Gastric emptying scintigraphy — Scintigraphy is performed to evaluate gastric emptying after eating a pancake labeled by 20 megabecquerel (MBq) Technetium-99m-Albumin (TC-99m-LyoMAA)
Other: Determination of gut hormones — Gut hormone levels will be determined after eating a standard meal in the RYGB and SG groups.
  Arms: Bad responder RYGB; Bad responder SG; Good responder RYGB; Good responder SG

SUMMARY:
The study evaluates the gastric emptying by scintigraphy in patients that had bariatric surgery (RYGB of gastric sleeve) comparing patients with successful and unsuccessful weight loss and in patients before and after the placement of a duodenal-jejunal bypass liner.

Additional, after bariatric surgery gut hormones that influence the gastric emptying rate are determined.

DETAILED DESCRIPTION:
Bariatric surgery reduces stomach volume and passage of foods through the gastrointestinal tract is altered. The satiety level often increases, which is probably caused by gut hormones. Patients response on different bariatric procedures varies widely and it is difficult to predict which patient responds well. Possibly, patients who have successful excess weight loss (EWL) two years after surgery have different gastric emptying rates compared to unsuccessful patients.

Changes in gut hormones after implantation of a duodenal-jejunal bypass liner were demonstrated in other studies. However, gastric emptying before and after placement of this liner is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to adhere to the study visit schedule and protocol requirements
* Patients must be able to give informed consent and the consent must be obtained prior to any study procedures
* Patients who had a follow-up period up till 2 years after bariatric surgery without any complications or
* Patients are eligible for DJBL implantation

Exclusion Criteria:

* Binge-eating or associated eating disorder
* Active drug or alcohol addiction
* Pregnancy or giving breast feeding
* Gluten allergy
* Inability to stop medication that affects the motility of the upper GI tract (anti-cholinergic drugs, prokinetics, theophylline, calcium blocking agents, opioids)
* Endocrine disease influencing gastric emptying (diabetes mellitus, hyper- or hypothyroidism). Type 2 diabetes mellitus is not an exclusion criterium for patients receiving the DJBL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Gastric emptying rate after bariatric surgery | 2 years after surgery
  In the RYGB and SG group
Change in gastric emptying rate after implantation of DJBL | before and 1 month after
  In the DJBL group

SECONDARY OUTCOMES:
Gut hormone levels after standard meal | 2 years after surgery
Weight loss after bariatric surgery | 2 years after bariatric surgery
Quality of life (SF-36, BAROS) after bariatric surgery | 2 years after bariatric surgery
Change in quality of life (SF-36, BAROS) after DJBL | Before and 1 month after implantation of DJBL

CONTACTS AND LOCATIONS:
Overall Officials: Frits J Berends, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate hospital, Arnhem, Netherlands

REFERENCES:
- [Background] Gersin KS, Keller JE, Stefanidis D, Simms CS, Abraham DD, Deal SE, Kuwada TS, Heniford BT. Duodenal- jejunal bypass sleeve: a totally endoscopic device for the treatment of morbid obesity. Surg Innov. 2007 Dec;14(4):275-8. doi: 10.1177/1553350607312901. PMID 18178916
- [Background] de Moura EG, Orso IR, Martins BC, Lopes GS, de Oliveira SL, Galvao-Neto Mdos P, Mancini MC, Santo MA, Sakai P, Ramos AC, Garrido-Junior AB, Halpern A, Cecconello I. Improvement of insulin resistance and reduction of cardiovascular risk among obese patients with type 2 diabetes with the duodenojejunal bypass liner. Obes Surg. 2011 Jul;21(7):941-7. doi: 10.1007/s11695-011-0387-0. PMID 21442376
- [Background] de Jonge C, Rensen SS, Verdam FJ, Vincent RP, Bloom SR, Buurman WA, le Roux CW, Schaper NC, Bouvy ND, Greve JW. Endoscopic duodenal-jejunal bypass liner rapidly improves type 2 diabetes. Obes Surg. 2013 Sep;23(9):1354-60. doi: 10.1007/s11695-013-0921-3. PMID 23526068
- [Background] Wang G, Agenor K, Pizot J, Kotler DP, Harel Y, Van Der Schueren BJ, Quercia I, McGinty J, Laferrere B. Accelerated gastric emptying but no carbohydrate malabsorption 1 year after gastric bypass surgery (GBP). Obes Surg. 2012 Aug;22(8):1263-7. doi: 10.1007/s11695-012-0656-6. PMID 22527599
- [Background] Dirksen C, Damgaard M, Bojsen-Moller KN, Jorgensen NB, Kielgast U, Jacobsen SH, Naver LS, Worm D, Holst JJ, Madsbad S, Hansen DL, Madsen JL. Fast pouch emptying, delayed small intestinal transit, and exaggerated gut hormone responses after Roux-en-Y gastric bypass. Neurogastroenterol Motil. 2013 Apr;25(4):346-e255. doi: 10.1111/nmo.12087. Epub 2013 Jan 29. PMID 23360316
- [Background] Braghetto I, Davanzo C, Korn O, Csendes A, Valladares H, Herrera E, Gonzalez P, Papapietro K. Scintigraphic evaluation of gastric emptying in obese patients submitted to sleeve gastrectomy compared to normal subjects. Obes Surg. 2009 Nov;19(11):1515-21. doi: 10.1007/s11695-009-9954-z. Epub 2009 Aug 28. PMID 19714384
- [Background] Melissas J, Daskalakis M, Koukouraki S, Askoxylakis I, Metaxari M, Dimitriadis E, Stathaki M, Papadakis JA. Sleeve gastrectomy-a "food limiting" operation. Obes Surg. 2008 Oct;18(10):1251-6. doi: 10.1007/s11695-008-9634-4. Epub 2008 Jul 29. PMID 18663545
- [Background] Baumann T, Kuesters S, Grueneberger J, Marjanovic G, Zimmermann L, Schaefer AO, Hopt UT, Langer M, Karcz WK. Time-resolved MRI after ingestion of liquids reveals motility changes after laparoscopic sleeve gastrectomy--preliminary results. Obes Surg. 2011 Jan;21(1):95-101. doi: 10.1007/s11695-010-0317-6. PMID 21088924
- [Background] Escalona A, Yanez R, Pimentel F, Galvao M, Ramos AC, Turiel D, Boza C, Awruch D, Gersin K, Ibanez L. Initial human experience with restrictive duodenal-jejunal bypass liner for treatment of morbid obesity. Surg Obes Relat Dis. 2010 Mar 4;6(2):126-31. doi: 10.1016/j.soard.2009.12.009. Epub 2010 Jan 20. PMID 20359665